CLINICAL TRIAL: NCT04166344
Title: Effectiveness of a Web-based, Digital Health Platform Combining Social Care and Respiratory Coach Support to Improve Adherence to Treatment and Symptom Control in Children and Adolescents with Difficult-to-control Asthma
Brief Title: A MHealth Intervention to Improve Symptom Control in Children and Adolescents with Difficult-to-control Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lovexair Foundation (Other)
Collaborators: Hospital Vall d'Hebron (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital Universitari Parc Salut Mar (Unknown); Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Raquel Sebio, Physiotherapist, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LVX-ASTHMA-2019
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Asthma in Children

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The statistical analyses will be performed by one researcher unaware of patient allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants in the IG will be given free access to the HappyAir platform during a 6-month period. This platform combines online/offline content to help patients with chronic respiratory diseases monitor their symptoms and improve self-management. In addition to tailored information on their condition, participants will be encouraged to fill in daily data on their physical activity levels, symptomatology, use of rescue medication and mood. In children under 12 years, parents or caregivers will fill in this information. Patients will be asked to record their peak expiratory flow using an electronic peak flow meter twice daily. Every patient will be assigned a respiratory coach who will monitor patient during the study and whom the patients can contact at any time.
  Interventions: Behavioral: Happyair Ecosystem
- Control Group (No Intervention): Subjects in the CG will receive standard care consisting of periodic visitations at the Allergology or Paediatric Pulmonology Unit in their respective hospitals every 4 - 8 weeks according to their physician's criteria. In addition, patients and caregivers in both groups will receive one educational session regarding the correct use of their inhalers.

INTERVENTIONS:
Behavioral: Happyair Ecosystem — Happyair Ecosystem is a Smart Community for the integral care of patients with chronic or rare respiratory diseases such as Asthma, COPD or Alfa-1.
  Our community provides online & offline training and resources in digital health and social care to patients, family, caregivers, healthcare professionals and researchers.
  Using our platform, all of our members will be able to connect in order to improve the health and well-being of patients, learn to manage self-care, ensure an active lifestyle, and contribute to the development of current and future research projects.
  Arms: Intervention Group

SUMMARY:
Asthma is the most common chronic respiratory disease worldwide. Despite advances in asthma management, control of the disease is still a challenge especially among children. Information and communications technology (ICT) have been recently used in clinical practice to increase awareness of diseases, encourage patients to engage in the management of their conditions and improve monitoring and surveillance. The investigators of this study will test a new digital platform combining online/offline content aimed to improve asthma control and reduce exacerbations and unnecessary consultations in children with difficult-to-control asthma. A randomised controlled trial enrolling 60 patients allocated in two groups has been designed. The intervention group (IG) will be granted free access during 6 months to a web-based platform. During this period, patient will have access to online/off line content to improve disease awareness, monitor signs and symptoms and will also get the support of a respiratory coach. In addition, patients in this group will receive an electronic peak flow meter to register daily variations in maximal expiratory flow and an electronic device to connect to their inhaler to track adequate intake of inhaled medication. The control group (CG) will receive usual care consisted of scheduled visitations to medical doctors every 4 - 8 weeks. Both groups will be evaluated at baseline, post-intervention (6 months) and at follow up (one year) in the following variables: age, gender, asthma severity classification according to international guidelines, date of diagnosis, weight, height, Body Mass Index (BMI), forced expiratory volume in 1 second (FEV1), Asthma Control Test (ACT) score, treatment received for asthma, number of exacerbations in the previous 6 months and concomitant diseases. Exacerbations will be defined as any worsening in asthma symptoms that requires an increase in the usual therapy, an unscheduled physician visit, treatment in the emergency room or hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* children between 6 and 18 years old;
* diagnosis of moderate to severe persistent asthma according to the international guidelines
* difficult to control asthma according to a scoring in the Asthma Control Questionnaire (ACQ) of 1.5 points or Asthma Control Test (ACT) ≤19;
* access to internet and a smartphone, tablet or computer;
* ability to understand and use the web-based platform (in children <12 years the ability of the tutor or legal guardian);
* informed consent (by the tutor or legal guardian)

Exclusion Criteria:

* patients who have had an exacerbation in the previous two weeks;
* patients with intermittent asthma and/or well-controlled asthma according to the Asthma Control Questionnaire (ACQ) score of <1.5 or Asthma Control Test (ACT) score ≥20;
* any neurological or psychiatric condition that prevents patients to use adequately the platform.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Differences in asthma control inter-group | 6 months
  Differences in asthma control (score) will be calculated according to the Asthma Control Test (ACT) in comparison with the control group. The ACT consists of five items that are rated according to a five-point scale where where 1 means poor control and 5 indicates better asthma control.
Differences in asthma control inter-group | 12 months
  Differences in asthma control (score) will be calculated according to the Asthma Control Test (ACT) in comparison with the control group. The ACT consists of five items that are rated according to a five-point scale where where 1 means poor control and 5 indicates better asthma control.

SECONDARY OUTCOMES:
Inclusion rates (feasibility) | Baseline
  Total number of patients recruited which consented from those eligible
Completion rates | 12 months
  Total number of patients who completed the interventions from those who were recruited
Incidence of exacerbations | 12 months
  Number of exacerbations (events) in a year in both groups. Exacerbations will be defined as any worsening in asthma symptoms that requires an increase in the usual therapy, an unscheduled physician visit, treatment in the emergency room or hospitalization.
Changes in lung function (FEV1) | 6 Months
  Lung function will be assessed by recording the Forced Expiratory Volume in the 1st second during a forced spirometry test.
Changes in lung function (FEV1) | 12 Months
  Lung function will be assessed by recording the Forced Expiratory Volume in the 1st second during a forced spirometry test.
Changes in lung function (PEF) | 6 Months
  Peak Expiratory flow will be recorded during a forced spirometry test to determine maximum expiratory flow as an indirect way of monitoring airway inflammation as well as asthma control over time.
Changes in lung function (PEF) | 12 Months
  Peak Expiratory flow will be recorded during a forced spirometry test to determine maximum expiratory flow as an indirect way of monitoring airway inflammation as well as asthma control over time.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitari Parc Taulí, Sabadell, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carvajal-Uruena I, Garcia-Marcos L, Busquets-Monge R, Morales Suarez-Varela M, Garcia de Andoin N, Batlles-Garrido J, Blanco-Quiros A, Lopez-Silvarrey A, Garcia-Hernandez G, Guillen-Grimaj F, Gonzalez-Diaz C, Bellido-Blasco J. [Geographic variation in the prevalence of asthma symptoms in Spanish children and adolescents. International Study of Asthma and Allergies in Childhood (ISAAC) Phase 3, Spain]. Arch Bronconeumol. 2005 Dec;41(12):659-66. doi: 10.1016/s1579-2129(06)60333-9. Spanish. PMID 16373042
- [Background] Sullivan PW, Ghushchyan V, Kavati A, Navaratnam P, Friedman HS, Ortiz B. Trends in Asthma Control, Treatment, Health Care Utilization, and Expenditures Among Children in the United States by Place of Residence: 2003-2014. J Allergy Clin Immunol Pract. 2019 Jul-Aug;7(6):1835-1842.e2. doi: 10.1016/j.jaip.2019.01.055. Epub 2019 Feb 15. PMID 30772478
- [Background] Morita PP, Yeung MS, Ferrone M, Taite AK, Madeley C, Stevens Lavigne A, To T, Lougheed MD, Gupta S, Day AG, Cafazzo JA, Licskai C. A Patient-Centered Mobile Health System That Supports Asthma Self-Management (breathe): Design, Development, and Utilization. JMIR Mhealth Uhealth. 2019 Jan 28;7(1):e10956. doi: 10.2196/10956. PMID 30688654
- [Background] Ahmed S, Ernst P, Bartlett SJ, Valois MF, Zaihra T, Pare G, Grad R, Eilayyan O, Perreault R, Tamblyn R. The Effectiveness of Web-Based Asthma Self-Management System, My Asthma Portal (MAP): A Pilot Randomized Controlled Trial. J Med Internet Res. 2016 Dec 1;18(12):e313. doi: 10.2196/jmir.5866. PMID 27908846
- [Background] van Gaalen JL, Beerthuizen T, van der Meer V, van Reisen P, Redelijkheid GW, Snoeck-Stroband JB, Sont JK; SMASHING Study Group. Long-term outcomes of internet-based self-management support in adults with asthma: randomized controlled trial. J Med Internet Res. 2013 Sep 12;15(9):e188. doi: 10.2196/jmir.2640. PMID 24028826
- [Background] Rasmussen LM, Phanareth K, Nolte H, Backer V. Internet-based monitoring of asthma: a long-term, randomized clinical study of 300 asthmatic subjects. J Allergy Clin Immunol. 2005 Jun;115(6):1137-42. doi: 10.1016/j.jaci.2005.03.030. PMID 15940125
- [Background] Barrett MA, Humblet O, Marcus JE, Henderson K, Smith T, Eid N, Sublett JW, Renda A, Nesbitt L, Van Sickle D, Stempel D, Sublett JL. Effect of a mobile health, sensor-driven asthma management platform on asthma control. Ann Allergy Asthma Immunol. 2017 Nov;119(5):415-421.e1. doi: 10.1016/j.anai.2017.08.002. PMID 29150069
- [Background] Newhouse N, Martin A, Jawad S, Yu LM, Davoudianfar M, Locock L, Ziebland S, Powell J. Randomised feasibility study of a novel experience-based internet intervention to support self-management in chronic asthma. BMJ Open. 2016 Dec 28;6(12):e013401. doi: 10.1136/bmjopen-2016-013401. PMID 28031210
- [Background] Christakis DA, Garrison MM, Lozano P, Meischke H, Zhou C, Zimmerman FJ. Improving parental adherence with asthma treatment guidelines: a randomized controlled trial of an interactive website. Acad Pediatr. 2012 Jul-Aug;12(4):302-11. doi: 10.1016/j.acap.2012.03.006. Epub 2012 Jun 11. PMID 22694878
- [Background] Reddel HK, Bateman ED, Becker A, Boulet LP, Cruz AA, Drazen JM, Haahtela T, Hurd SS, Inoue H, de Jongste JC, Lemanske RF Jr, Levy ML, O'Byrne PM, Paggiaro P, Pedersen SE, Pizzichini E, Soto-Quiroz M, Szefler SJ, Wong GW, FitzGerald JM. A summary of the new GINA strategy: a roadmap to asthma control. Eur Respir J. 2015 Sep;46(3):622-39. doi: 10.1183/13993003.00853-2015. Epub 2015 Jul 23. PMID 26206872
- [Background] Sastre J, Olaguibel J, Vega JM, Del Pozo V, Picado C, Lopez Vina A. Cut-off points for defining asthma control in three versions of the Asthma Control Questionnaire. J Asthma. 2010 Oct;47(8):865-70. doi: 10.3109/02770903.2010.491149. PMID 20846084
- [Background] Juniper EF, Gruffydd-Jones K, Ward S, Svensson K. Asthma Control Questionnaire in children: validation, measurement properties, interpretation. Eur Respir J. 2010 Dec;36(6):1410-6. doi: 10.1183/09031936.00117509. Epub 2010 Jun 7. PMID 20530041
- [Background] Picado C, Badiola C, Perulero N, Sastre J, Olaguibel JM, Lopez Vina A, Vega JM; Covalair Investigator Group. Validation of the Spanish version of the Asthma Control Questionnaire. Clin Ther. 2008 Oct;30(10):1918-31. doi: 10.1016/j.clinthera.2008.10.005. PMID 19014848